CLINICAL TRIAL: NCT03741114
Title: Intrauterine Inflated Foley's Catheter Balloon Plus Intravenous Tranexamic Acid During Cesarean Delivery for Complete Placenta Previa: a Randomized Double-blind Controlled Trial
Brief Title: Foley's Catheter Balloon Plus Tranexamic Acid During Cesarean Delivery for Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/199/18
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Placenta Previa
Keywords: placenta previa; tranexamic acid; cesarean section; Foley's Catheter Balloon
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: The study was a double-blind randomized controlled trial carried out in a tertiary University Hospital
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which was used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley's Catheter plus TA (Active Comparator): patients managed by Intrauterine Inflated Foley's Catheter Balloon after delivery of the fetus plus 1 gm tranexamic acid in 100ml saline intravenous just before skin incision
  Interventions: Procedure: Foley's Catheter; Drug: TA
- Foley's Catheter plus placebo to TA (Active Comparator): patients managed by Intrauterine Inflated Foley's Catheter Balloon after delivery of the fetus plus single injection of 100 ml intravenous saline before skin incision
  Interventions: Procedure: Foley's Catheter; Drug: Placebo

INTERVENTIONS:
Procedure: Foley's Catheter — patients managed by Intrauterine Inflated Foley's Catheter Balloon after delivery of the fetus.
  Other Names: Active Comparator
Drug: TA — patients received 1 gm tranexamic acid intravenous just before skin incision in 100 ml saline
  Other Names: active comparator
  Arms: Foley's Catheter plus TA
Drug: Placebo — patients received 100 ml saline just before skin incision
  Other Names: Placebo to TA
  Arms: Foley's Catheter plus placebo to TA

SUMMARY:
Placenta previa (PP) is an obstetric condition that is closely linked with massive obstetric hemorrhage with a varied incidence about once in every 150-250 live births. Insertion of intrauterine balloon tamponade has been suggested in the management of massive postpartum hemorrhage (PPH). The Bakri balloon has a sausage-like spindle shape and a drainage lumen and is made of silicon. It has been used in cases of uterine atony and placenta previa with a success rate of 90%. However, Bakri balloon is not available in all countries.

The aim of this study is to evaluate the efficacy of the use of intrauterine inflated Foley's catheter balloon with or without intravenous tranexamic acid to control PPH during cesarean delivery in cases of placenta previa.

DETAILED DESCRIPTION:
Eligible participants were allocated to one of two groups. Group (I): patients managed by Intrauterine Inflated Foley's Catheter Balloon after delivery of the fetus. Group (II): patients received 1 gm tranexamic acid (TA), (2 ampoules of Capron® 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision plus Intrauterine Inflated Foley's Catheter Balloon. In group I, patients received a single injection of intravenous saline before skin incision prepared in a syringe and coded by a pharmacist in the pharmacy of the hospital. Neither the surgeon nor the anesthetist will know the nature of the IV administered drug before cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single term fetus scheduled for an elective cesarean section for complete placenta previa

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease
* patients with the high possibility of the morbid adherent placenta
* known coagulopathy or thromboembolic disease
* those presented with severe antepartum hemorrhage
* hypersensitivity or contraindications of use of tranexamic acid
* patient refuses to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All pregnant women with a single term fetus scheduled for an elective cesarean section for complete placenta previa
Enrollment: 120 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 24 hours post operative
  number of participant with blood loss > 1000ml

SECONDARY OUTCOMES:
intraoperative blood loss | during the operation
  amount of blood loss during cesarean section
The number of participant needed for blood transfusion | 24 hours postoperative
  Calculation of the number of participant needed for blood transfusion
number of participant need of extra surgical maneuvers | 24 hours post operative
  number of participant need of extra surgical maneuvers like internal iliac ligation or hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided